CLINICAL TRIAL: NCT02891252
Title: Randomized Investigation of Thyroid Operation as Day Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJ-495
Record Dates: First submitted 2016-09-01; First posted 2016-09-07 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-05

CONDITIONS: Hemithyroidectomy; Outpatient; Hemmorhage
MeSH Terms: interventions — Ambulatory Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- outpatient (Active Comparator): outpatient
  Interventions: Procedure: outpatient procedure
- inpatient (No Intervention): inpatient

INTERVENTIONS:
Procedure: outpatient procedure
  Arms: outpatient

SUMMARY:
hemithyroidectomy as a outpatient procedure is performed in some countries, it has never been done a RCT whether it is feasible

DETAILED DESCRIPTION:
Many surgical procedures, which previously resulted in days to week's hospital admissions, are now done as outpatient procedures. This is the result of better surgical and anaesthesiology techniques as well as the economic incentive.

Examples from another surgical fields are cholecystectomy and further back in oto-rhino- laryngology (ORL) also tonsillectomy.

Hemithyriodectomy as an outpatient procedure is becoming increasingly popular and is already applied in some countries. However many European countries is continuing the procedure with hospital admission post-operatively (inpatient surgery), due to risk of complications. In Denmark hemithyroidectomy is currently done with at least one night hospital admission for observation of above mentioned . At the ORL department at Køge hospital it is annually performed approximately 200 hemithyroidectomies. It is a common procedure and the number of procedures yearly is increasing. Complications to hemithyroidectomy include postoperative haemorrhage, damage to the recurrent laryngeal nerve, hypothyroidism and infection and veryn rarely hypocalcaemia. With sufficient patient information, the above-mentioned complications can be managed in an outpatient setting. Postoperative haemorrhage is the most serious complication and thyroid surgery is unique in outpatient setting, considering the risk of cervical haemorrhage which secondary can lead to respiratory failure due to tracheal compression and laryngeal oedema in a rapid sequence. Incidence of haemorrhage after thyroid surgery varies from 0.19 % to 2.8 % of which most bleedings occur within six hours postoperatively. There are two different approaches in the event of post- operative haemorrhage; acute decompression bedside and acute re-operation.

Acute decompression is reserved for respiratory failures. Eligibility criteria for who may undergo outpatient thyroid surgery have been debated in the literature. No consensus has been reached for these criteria. For now, there is consensus that some patients (high risk of bleeding) will require inpatient procedure, and in carefully selected groups of patients outpatient thyroid surgery is already performed, as the inclusion criteria below. Outpatient hemithyroidectomy has shown low number of complications in retrospective studies as well as high patient acceptance and economical advantage in recent prospective and retrospective studies studies. However, recent national and international studies recommend against outpatient procedure, mainly due to the risk of late cervical haemorrhage. It is therefore important to continue to investigate whether hemithyroidectomyis feasible as an outpatient procedure, especially considering patient safety and acceptance. This will be done in a randomized controlled trial where half of the patients are allocated to outpatient procedure and the other half to inpatient procedure. The aim is non-inferiority comparing the two above-mentioned procedures. As far as the authors know, no previous RCT has been done or published with this purpose.

ELIGIBILITY:
Inclusion Criteria:

The hospitals normal outpatient criteria (ASA II or I), adult person to stay

with patient on night of surgery) Euthyroid Normal function of vocal cords preoperatively Lives within a 30 km radius or within 45 minutes away with ambulance, from the hospital Speaks Danish

Exclusion Criteria:

Suspected malignancy Previous thyroid or major neck surgery Intrathoracic thyroid gland Former treatment with radioactive iodine Anticoagulation treatment except ASA and ADP inhibitors

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients that are converted to inpatient and/or re- admitted within 24h are under 20% in the outpatient group | 24 h

SECONDARY OUTCOMES:
Patient acceptance to outpatient procedure from patient satisfactory questionnaire (Appendix 1). | 4 weeks
Difference in postoperative haemorrhage | 24 h
Difference in mean level of NRS pain scores at rest based on measurements at 2h and 20h on POD0 and at 8h and 20 h on POD 1. | 24 h
Difference in mean level of NRS pain scores during swallowing of saliva based on measurements at 2h and 20h on POD0 and at 8h and 20 h on POD 1. | 24 h
Difference in mean levels of NRS nausea at 2h, 20h (POD 0) and at 8h and 20h (POD1) | 24 h
Difference in NRS rated quality of sleep and level of tiredness at 8h on POD1 | 24 h

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen University Hospital, Køge, Denmark

IPD SHARING:
Plan to Share IPD: Yes
v

REFERENCES:
- [Derived] Haugaard CF, Homoe P, Nygren A, Mathiesen O, Hansen LN, Hvilsom GB. Randomised controlled trial of in- versus out-patient management of benign hemithyroidectomy. Dan Med J. 2023 Dec 6;71(1):A06230377. PMID 38235985